CLINICAL TRIAL: NCT02153307
Title: Ambulatory Electrocardiographic Monitoring for the Detection of High-Degree Atrio-Ventricular Block in Patients With New-onset PeRsistent LEft Bundle Branch Block After Transcatheter Aortic Valve Implantation. The "MARE" Study
Acronym: MARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MARE
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Aortic Valve Disease; Conduction Disturbances
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable loop recorders Reveal ICM LINQ®, (Experimental)
  Interventions: Device: Implantable loop recorders system Reveal ICM LINQ®,

INTERVENTIONS:
Device: Implantable loop recorders system Reveal ICM LINQ®,

SUMMARY:
The purpose of this study is to determine the incidence and predictors of high degree or complete atrioventricular block (AVB) (paroxysmal or persistent) in patients with new-onset persistent left bundle branch block (NOP-LBBB) following transcatheter aortic valve implantation (TAVI) and to evaluate the usefulness of the Reveal LINQ® insertable Cardiac Monitor (ICM) (Medtronic, Inc., Minneapolis, USA) for the detection of significant arrhythmias in patients with NOP-LBBB following TAVI.

DETAILED DESCRIPTION:
This is a prospective observational study including patients undergoing TAVI with either self- or balloon-expandable valves. After the procedure, patients will be on ECG monitoring during the hospitalization period (or at least 72 hours), and an ECG will be performed daily until hospital discharge in all patients. Patients with new-onset persistent LBBB at hospital discharge (new-onset LBBB of a duration of at least 48 h which persists at hospital discharge, at least 3 days and up to 15 days after the procedure) will receive an implantable loop recorder Reveal ICM LINQ®, which will be implanted subcutaneously to record adequate QRS complexes and P waves. The patients will be followed in outpatient clinic visits at 1, 12, 24 and 36 months after TAVR, or if symptoms suggestive of cardiac origin or relevant arrhythmic events occur. The device will be manually interrogated in each visit. Phone contacts will be also carried out every three months.

ELIGIBILITY:
Inclusion Criteria:

-Patients undergoing TAVI with either balloon or self-expandable valves who develop new-onset LBBB persistent at hospital discharge, at least 3 days after the procedure

Exclusion Criteria:

* Failure to provide informed consent
* Baseline pacemaker/defibrillator or pacemaker/defibrillator implanted during the hospitalization period following the TAVI procedure
* Pre-existing complete LBBB
* Patients with a life-expectancy of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-05 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
-Rate and time of onset of high degree or complete AVB | 1Year
-Incidence of arrhythmic events identified by the IRL leading to a change in treatment or major adverse event | 1 Year

SECONDARY OUTCOMES:
-Rate of high degree or complete of AVB | Within the first month after TAVI procedure
-Rate of high degree or complete of AVB | 6-month follow-up
-Rate of high degree or complete AVB | 24-month follow-up
-Rate of high degree or complete AVB | 36-month follow-up
-Electrocardiographic and device-related factors predicting the occurence of high degree or complete AVB in patients with new-onset LBBB after TAVI | Within the first 3 years following TAVI procedure
  Periprocedural results of TAVI of patients with NOP-LVV will be used to characterize predictors of high degree or complete AVB. Moreover, electrocardiographic characteristics at hospital discharge of patients with NOP-LVV will also be used to characterize predictors of high degree or complete AVB.
-Rate of new atrial fibrillation or ventricular arrhythmias | Within the first 3 years following TAVI procedure
-Changes in left ventricular function and mitral regurgitation over time | Within the first 3 years following TAVI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes, MD, Principal Investigator — Fondation IUCPQ
Locations (1):
- IUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Background] Piazza N, de Jaegere P, Schultz C, Becker AE, Serruys PW, Anderson RH. Anatomy of the aortic valvar complex and its implications for transcatheter implantation of the aortic valve. Circ Cardiovasc Interv. 2008 Aug;1(1):74-81. doi: 10.1161/CIRCINTERVENTIONS.108.780858. PMID 20031657
- [Background] Thompson R, Mitchell A, Ahmed M, Towers M, Yacoub M. Conduction defects in aortic valve disease. Am Heart J. 1979 Jul;98(1):3-10. doi: 10.1016/0002-8703(79)90313-2. No abstract available. PMID 313146
- [Background] El-Khally Z, Thibault B, Staniloae C, Theroux P, Dubuc M, Roy D, Guerra P, Macle L, Talajic M. Prognostic significance of newly acquired bundle branch block after aortic valve replacement. Am J Cardiol. 2004 Oct 15;94(8):1008-11. doi: 10.1016/j.amjcard.2004.06.055. PMID 15476613
- [Background] Thomas JL, Dickstein RA, Parker FB Jr, Potts JL, Poirier RA, Fruehan CT, Eich RH. Prognostic significance of the development of left bundle conduction defects following aortic valve replacement. J Thorac Cardiovasc Surg. 1982 Sep;84(3):382-6. PMID 7109669
- [Background] Foppl M, Hoffmann A, Amann FW, Roth J, Stulz P, Hasse J, Gradel E, Burckhardt D. Sudden cardiac death after aortic valve surgery: incidence and concomitant factors. Clin Cardiol. 1989 Apr;12(4):202-7. doi: 10.1002/clc.4960120405. PMID 2714032
- [Background] van der Boon RM, Nuis RJ, Van Mieghem NM, Jordaens L, Rodes-Cabau J, van Domburg RT, Serruys PW, Anderson RH, de Jaegere PP. New conduction abnormalities after TAVI--frequency and causes. Nat Rev Cardiol. 2012 May 1;9(8):454-63. doi: 10.1038/nrcardio.2012.58. PMID 22547171
- [Background] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for Transcatheter Aortic Valve Implantation clinical trials: a consensus report from the Valve Academic Research Consortium. J Am Coll Cardiol. 2011 Jan 18;57(3):253-69. doi: 10.1016/j.jacc.2010.12.005. Epub 2011 Jan 7. PMID 21216553
- [Background] Dou J, Xia L, Zhang Y, Shou G, Wei Q, Liu F, Crozier S. Mechanical analysis of congestive heart failure caused by bundle branch block based on an electromechanical canine heart model. Phys Med Biol. 2009 Jan 21;54(2):353-71. doi: 10.1088/0031-9155/54/2/012. Epub 2008 Dec 19. PMID 19098354
- [Background] Piazza N, Nuis RJ, Tzikas A, Otten A, Onuma Y, Garcia-Garcia H, Schultz C, van Domburg R, van Es GA, van Geuns R, de Jaegere P, Serruys PW. Persistent conduction abnormalities and requirements for pacemaking six months after transcatheter aortic valve implantation. EuroIntervention. 2010 Sep;6(4):475-84. doi: 10.4244/EIJ30V6I4A80. PMID 20884435
- [Background] Houthuizen P, Van Garsse LA, Poels TT, de Jaegere P, van der Boon RM, Swinkels BM, Ten Berg JM, van der Kley F, Schalij MJ, Baan J Jr, Cocchieri R, Brueren GR, van Straten AH, den Heijer P, Bentala M, van Ommen V, Kluin J, Stella PR, Prins MH, Maessen JG, Prinzen FW. Left bundle-branch block induced by transcatheter aortic valve implantation increases risk of death. Circulation. 2012 Aug 7;126(6):720-8. doi: 10.1161/CIRCULATIONAHA.112.101055. Epub 2012 Jul 12. PMID 22791865
- [Background] Testa L, Latib A, De Marco F, De Carlo M, Agnifili M, Latini RA, Petronio AS, Ettori F, Poli A, De Servi S, Ramondo A, Napodano M, Klugmann S, Ussia GP, Tamburino C, Brambilla N, Colombo A, Bedogni F. Clinical impact of persistent left bundle-branch block after transcatheter aortic valve implantation with CoreValve Revalving System. Circulation. 2013 Mar 26;127(12):1300-7. doi: 10.1161/CIRCULATIONAHA.112.001099. Epub 2013 Feb 26. PMID 23443735
- [Background] Urena M, Mok M, Serra V, Dumont E, Nombela-Franco L, DeLarochelliere R, Doyle D, Igual A, Larose E, Amat-Santos I, Cote M, Cuellar H, Pibarot P, de Jaegere P, Philippon F, Garcia del Blanco B, Rodes-Cabau J. Predictive factors and long-term clinical consequences of persistent left bundle branch block following transcatheter aortic valve implantation with a balloon-expandable valve. J Am Coll Cardiol. 2012 Oct 30;60(18):1743-52. doi: 10.1016/j.jacc.2012.07.035. Epub 2012 Oct 3. PMID 23040577
- [Background] Moya A, Garcia-Civera R, Croci F, Menozzi C, Brugada J, Ammirati F, Del Rosso A, Bellver-Navarro A, Garcia-Sacristan J, Bortnik M, Mont L, Ruiz-Granell R, Navarro X; Bradycardia detection in Bundle Branch Block (B4) study. Diagnosis, management, and outcomes of patients with syncope and bundle branch block. Eur Heart J. 2011 Jun;32(12):1535-41. doi: 10.1093/eurheartj/ehr071. Epub 2011 Mar 28. PMID 21444367
- [Background] Krahn AD, Klein GJ, Yee R, Takle-Newhouse T, Norris C. Use of an extended monitoring strategy in patients with problematic syncope. Reveal Investigators. Circulation. 1999 Jan 26;99(3):406-10. doi: 10.1161/01.cir.99.3.406. PMID 9918528
- [Background] Lombardi F, Calosso E, Mascioli G, Marangoni E, Donato A, Rossi S, Pala M, Foti F, Lunati M. Utility of implantable loop recorder (Reveal Plus) in the diagnosis of unexplained syncope. Europace. 2005 Jan;7(1):19-24. doi: 10.1016/j.eupc.2004.09.003. PMID 15670962
- [Background] Furukawa T, Maggi R, Bertolone C, Fontana D, Brignole M. Additional diagnostic value of very prolonged observation by implantable loop recorder in patients with unexplained syncope. J Cardiovasc Electrophysiol. 2012 Jan;23(1):67-71. doi: 10.1111/j.1540-8167.2011.02133.x. Epub 2011 Jul 21. PMID 21777327
- [Background] Paruchuri V, Adhaduk M, Garikipati NV, Steinberg JS, Mittal S. Clinical utility of a novel wireless implantable loop recorder in the evaluation of patients with unexplained syncope. Heart Rhythm. 2011 Jun;8(6):858-63. doi: 10.1016/j.hrthm.2011.01.039. Epub 2011 Feb 2. PMID 21296683
- [Background] Krahn AD, Klein GJ, Yee R, Hoch JS, Skanes AC. Cost implications of testing strategy in patients with syncope: randomized assessment of syncope trial. J Am Coll Cardiol. 2003 Aug 6;42(3):495-501. doi: 10.1016/s0735-1097(03)00659-4. PMID 12906979
- [Background] Task Force members; Brignole M, Vardas P, Hoffman E, Huikuri H, Moya A, Ricci R, Sulke N, Wieling W; EHRA Scientific Documents Committee; Auricchio A, Lip GY, Almendral J, Kirchhof P, Aliot E, Gasparini M, Braunschweig F; Document Reviewers; Lip GY, Almendral J, Kirchhof P, Botto GL; EHRA Scientific Documents Committee. Indications for the use of diagnostic implantable and external ECG loop recorders. Europace. 2009 May;11(5):671-87. doi: 10.1093/europace/eup097. No abstract available. PMID 19401342
- [Background] Crossley GH, Boyle A, Vitense H, Chang Y, Mead RH; CONNECT Investigators. The CONNECT (Clinical Evaluation of Remote Notification to Reduce Time to Clinical Decision) trial: the value of wireless remote monitoring with automatic clinician alerts. J Am Coll Cardiol. 2011 Mar 8;57(10):1181-9. doi: 10.1016/j.jacc.2010.12.012. Epub 2011 Jan 20. PMID 21255955
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738
- [Background] Surawicz B, Childers R, Deal BJ, Gettes LS, Bailey JJ, Gorgels A, Hancock EW, Josephson M, Kligfield P, Kors JA, Macfarlane P, Mason JW, Mirvis DM, Okin P, Pahlm O, Rautaharju PM, van Herpen G, Wagner GS, Wellens H; American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; American College of Cardiology Foundation; Heart Rhythm Society. AHA/ACCF/HRS recommendations for the standardization and interpretation of the electrocardiogram: part III: intraventricular conduction disturbances: a scientific statement from the American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; the American College of Cardiology Foundation; and the Heart Rhythm Society. Endorsed by the International Society for Computerized Electrocardiology. J Am Coll Cardiol. 2009 Mar 17;53(11):976-81. doi: 10.1016/j.jacc.2008.12.013. No abstract available. PMID 19281930
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Heart Rhythm Society. 2012 ACCF/AHA/HRS focused update incorporated into the ACCF/AHA/HRS 2008 guidelines for device-based therapy of cardiac rhythm abnormalities: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. Circulation. 2013 Jan 22;127(3):e283-352. doi: 10.1161/CIR.0b013e318276ce9b. Epub 2012 Dec 19. No abstract available. PMID 23255456
- [Background] Goldberger JJ, Cain ME, Hohnloser SH, Kadish AH, Knight BP, Lauer MS, Maron BJ, Page RL, Passman RS, Siscovick D, Siscovick D, Stevenson WG, Zipes DP; American Heart Association; American College of Cardiology Foundation; Heart Rhythm Society. American Heart Association/American College of Cardiology Foundation/Heart Rhythm Society scientific statement on noninvasive risk stratification techniques for identifying patients at risk for sudden cardiac death: a scientific statement from the American Heart Association Council on Clinical Cardiology Committee on Electrocardiography and Arrhythmias and Council on Epidemiology and Prevention. Circulation. 2008 Sep 30;118(14):1497-1518. No abstract available. PMID 18833586
- [Derived] Muntane-Carol G, Urena M, Nombela-Franco L, Amat-Santos I, Kleiman N, Munoz-Garcia A, Atienza F, Serra V, Deyell MW, Veiga-Fernandez G, Masson JB, Canadas-Godoy V, Himbert D, Castrodeza J, Elizaga J, Francisco Pascual J, Webb JG, de la Torre Hernandez JM, Asmarats L, Pelletier-Beaumont E, Philippon F, Rodes-Cabau J. Arrhythmic burden in patients with new-onset persistent left bundle branch block after transcatheter aortic valve replacement: 2-year results of the MARE study. Europace. 2021 Feb 5;23(2):254-263. doi: 10.1093/europace/euaa213. PMID 33083813
- [Derived] Rodes-Cabau J, Urena M, Nombela-Franco L, Amat-Santos I, Kleiman N, Munoz-Garcia A, Atienza F, Serra V, Deyell MW, Veiga-Fernandez G, Masson JB, Canadas-Godoy V, Himbert D, Castrodeza J, Elizaga J, Francisco Pascual J, Webb JG, de la Torre JM, Asmarats L, Pelletier-Beaumont E, Philippon F. Arrhythmic Burden as Determined by Ambulatory Continuous Cardiac Monitoring in Patients With New-Onset Persistent Left Bundle Branch Block Following Transcatheter Aortic Valve Replacement: The MARE Study. JACC Cardiovasc Interv. 2018 Aug 13;11(15):1495-1505. doi: 10.1016/j.jcin.2018.04.016. Epub 2018 Jul 18. PMID 30031719